CLINICAL TRIAL: NCT03333668
Title: Experimental fMRI Study on the Comparison of the Brain Function Effects of a Single Dose of Guanfacine and Lisdexamfetamine Relative to Placebo in Children and Adolescents With ADHD.
Brief Title: Experimental fMRI Study of Guanfacine and Lisdexamfetamine in ADHD Adolescents
Acronym: AGUALIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PCCWUAR
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: ADHD
Keywords: Lisdexamfetamine; Guanfacine; functional Magnetic Resonance Imaging; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Guanfacine

STUDY DESIGN:
Intervention Model Description: Each participant will complete all three experimental conditions (LISDEX, GXR, placebo) in a randomised order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lisdexamfetamine - Placebo (Active Comparator)
  Interventions: Drug: Lisdexamfetamine dimesylate; Drug: Placebo
- Guanfacine - Placebo (Active Comparator)
  Interventions: Drug: Guanfacine Extended Release Oral Tablet; Drug: Placebo
- Lisdexamfetamine - Guanfacine (Experimental)
  Interventions: Drug: Lisdexamfetamine dimesylate; Drug: Guanfacine Extended Release Oral Tablet

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — Lisdexamfetamine dimesylate (30mg for smaller, 50mg for larger boys) tablet
  Other Names: Vyvanse (Shire Pharmaceuticals Ltd.)
  Arms: Lisdexamfetamine - Guanfacine; Lisdexamfetamine - Placebo
Drug: Guanfacine Extended Release Oral Tablet — Guanfacine Extended Release (0.05mg/kg) tablet
  Other Names: Intuniv (Shire Pharmaceuticals Ltd.)
  Arms: Guanfacine - Placebo; Lisdexamfetamine - Guanfacine
Drug: Placebo — Vitamin C (10mg) tablet
  Arms: Guanfacine - Placebo; Lisdexamfetamine - Placebo

SUMMARY:
This is not a clinical trial. The aim of this study is to understand the mechanism of action of two recently licensed drugs for ADHD on brain function. We will compare the brain activation changes elicited by Guanfacine extended release (GXR; a non-stimulant drug) with the brain activation changes elicited by Lisdexamfetamine (LISDEX; a stimulant drug) and by placebo in 20 drug-free patients with ADHD using functional Magnetic Resonance Imaging (fMRI). For this purpose we intend to scan participants during their performance of tasks of attention, working memory, and inhibition, which we know from previous studies to elicit abnormal brain activation patterns in ADHD patients (Rubia et al., 2005; Smith et al., 2006).

DETAILED DESCRIPTION:
Twenty ADHD patients between 8 and 20 years of age will participate in the double-blind, randomised, active drug condition, within-group, placebo-controlled experimental fMRI study. Each participant will be assessed in baseline measures during a pre-assessment visit. Then the patient will be scanned 3 times under each of these 3 drug conditions: GXR, LISDEX, and placebo. Every patient will receive a single typical clinical weight-adjusted dose of GXR (0.05mg/kg rounded down to the closest dose of 1mg, 2mg, or a maximum of 3mg), LISDEX (for participants aged 8-9 years 20mg regardless of weight; for participants aged 10-20 years the dose will be calculated at 0.5mg/kg rounded to the closest 30, 40, or 50mg, middle doses, e.g. 35mg, will be rounded down) and placebo (10mg Vit C) in one of the scans, in a randomised order. Patients will perform a battery of cognitive tests 3.5 hours after drug administration, after which the will undergo an fMRI scan. The scan will start 4.5 hours after drug administration where drugs have shown to have maximum plasma concentration. Participants will be scanned 3 times, one week apart, under each drug condition.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 8-20 years
* Medication-naïve or non-medicated for two weeks or on stimulant medication, and willing to take the medication off for 48 hours before scans.
* Meeting DSM-5 diagnosis of ADHD
* Score above clinical cut-off on the ADHD module of the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) (Kaufman et al., 1997)
* Score above clinical cut-off for ADHD on the short forms of the Conners Parent Rating Scales, CPRS (Conners et al., 2008)
* Score above cut-off on the ADHD Rating Scale, ADHD-RS (DuPaul, et al., 1998)
* IQ > 70 as tested on the WASI-II (Wechsler et al., 1999)
* Mood and depression symptoms will be allowed as long as they are not the primary diagnosis.

Exclusion Criteria:

* IQ < 70 (Wechsler et al., 1999).
* Comorbidity with schizophrenia, bipolar disorder, learning disability, OCD, severe depression with current suicidal behaviour (as assessed by a clinical interview)
* Neurological problems, i.e. a history of severe neurological illness, e.g. brain tumour, epilepsy or a history of symptomatic seizures, polyneuropathy etc.
* Substance abuse history
* Other illness (cardiovascular, renal, hepatic, metabolic) that would impact the data integrity or safety of the subject (i.e. contraindicated to any of the treatments) as determined by the investigators
* Contraindication to MRI. i.e., previous implantation of metallic material, pacemaker, implanted medication pumps, neural stimulators, claustrophobia
* Unable to give informed assent or consent in the case of the parent
* Contraindications for LISDEX and GXR use (i.e. advanced arteriosclerosis, agitated states, hyperexcitability, hyperthyroidism, moderate or severe hypertension, symptomatic cardiovascular disease)

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in brain activation under the three drug conditions (LISDEX, GXR, placebo) | 2 weeks (3 hourly scans one week apart)
  Brain activation as measured by blood-oxygen-level-dependent (BOLD) response obtained by fMRI for each of the 3 below listed tasks and functional connectivity measures for the resting state scan.
  1. A working memory task (N-back)
  2. A tracking stop task
  3. A parametric sustained attention task

SECONDARY OUTCOMES:
Changes in dependent variables extracted from performance on the fMRI tasks used under the three drug conditions (LISDEX, GXR, placebo) | 2 weeks (3 hourly scans one week apart)
  1. A working memory task (N-back)
  2. A tracking stop task
  3. A parametric sustained attention task
Changes in dependent variables extracted from performance on a task battery outside the MRI scanner | 2 weeks (3 sessions one week apart)
  Gonogo task, Simon task, Continuous performance task, Vigilance task, Time Discrimination task

CONTACTS AND LOCATIONS:
Overall Officials: Katya Rubia, PhD, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology & Neuroscience; King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rubia K, Smith AB, Brammer MJ, Toone B, Taylor E. Abnormal brain activation during inhibition and error detection in medication-naive adolescents with ADHD. Am J Psychiatry. 2005 Jun;162(6):1067-75. doi: 10.1176/appi.ajp.162.6.1067. PMID 15930054
- [Background] Smith AB, Taylor E, Brammer M, Toone B, Rubia K. Task-specific hypoactivation in prefrontal and temporoparietal brain regions during motor inhibition and task switching in medication-naive children and adolescents with attention deficit hyperactivity disorder. Am J Psychiatry. 2006 Jun;163(6):1044-51. doi: 10.1176/ajp.2006.163.6.1044. PMID 16741205
- [Derived] El Masri S, Kowalczyk OS, Chiu TH, Criaud M, Lukito S, Mazibuko N, Salazar de Pablo G, Perez Rodriguez V, Makos O, Lam SL, Westwood S, Eaton-Turner A, Bozhilova N, Conti A, Santosh P, Roessner V, Kohls G, Mehta MA, Rubia K. Differential effects of a single dose of Lisdexamfetamine and Guanfacine on cognitive function in children with ADHD. Front Psychiatry. 2025 Nov 3;16:1676472. doi: 10.3389/fpsyt.2025.1676472. eCollection 2025. PMID 41256939

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03333668/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03333668/ICF_001.pdf